CLINICAL TRIAL: NCT02069314
Title: Diet and Muscle Function In Older Adults
Acronym: S32
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Professor, Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 1203012093
Record Dates: First submitted 2014-02-12; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2013-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Carbohydrates; Glucans; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whey protein supplementation (Experimental): 50 grams of whey blended into frozen drink
  Interventions: Dietary Supplement: Whey protein supplementation
- Carbohydrate supplementation (Experimental): 50 grams of polycose blended into frozen drink
  Interventions: Dietary Supplement: Carbohydrate (polycose) supplementation

INTERVENTIONS:
Dietary Supplement: Whey protein supplementation — subjects are asked to consume a smoothie with whey protein added
  Arms: Whey protein supplementation
Dietary Supplement: Carbohydrate (polycose) supplementation — Subjects are asked to consume a beverage with polycose added
  Arms: Carbohydrate supplementation

SUMMARY:
This research study was conducted to investigate the effects of a high protein diet on the efficiency of energy use at rest and at low-levels of physical activity. The hypothesis was that a high intake of dietary protein would result in a less efficient use of energy in skeletal muscle in older adults.

DETAILED DESCRIPTION:
This research study was conducted to investigate the effects of a high protein diet on the efficiency of energy use at rest and at low-levels of physical activity. The hypothesis was that a high intake of dietary protein would result in a less efficient use of energy in skeletal muscle in older adult

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older

Exclusion Criteria:

* Diabetic
* Acute symptoms of cardiovascular disease or congestive heart failure
* uncontrolled hypertension
* supplemental oxygen consumption at rest or during exercise
* lactose intolerance
* inability to ride a stationary cycle

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Dietary protein effects on muscle energy use | participants will be measured over an average of 26 days
  gross mechanical efficiency of muscle, consuming high and low protein supplements

SECONDARY OUTCOMES:
Effect of protein supplements on food intake | participants will be measured over an average of 26 days
  effects of high protein or high carbohydrate supplements on overall energy consumption in older adults.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, Ph.D., Principal Investigator — Purdue University Dept of Nutrition Science
Locations (1):
- Purdue University, West Lafayette, Indiana, United States